CLINICAL TRIAL: NCT02475616
Title: A Randomized, Double-blind, Single Ascending Oral Dose Study To Evaluate Safety, Tolerability And Pharmacokinetics Of PCO371 In Healthy Volunteers
Brief Title: A Single Ascending Dose Study of PCO371 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCO001US
Record Dates: First submitted 2015-06-02; First posted 2015-06-19 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
MeSH Terms: interventions — PCO371

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PCO371 (Experimental): Single oral dose of PCO371
  Interventions: Drug: PCO371
- Placebo Comparator (Placebo Comparator): Single oral dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PCO371
  Arms: PCO371
Drug: Placebo
  Arms: Placebo Comparator

SUMMARY:
This is a single-center, placebo-controlled, randomized, double-blind, dose-escalation study to evaluate safety, tolerability, and PK of a single oral (PO) administration of PCO371 in healthy adult males.

Caucasian and Japanese subjects will be randomized to receive either PCO371 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 45 years.
* Caucasian(BMI 18-30 mg/kg2) or first generation japanese(BMI 18-25kg/m2)
* Able and willing to abide by the protocol

Exclusion Criteria:

* Evidence of any medical condition that could affect renal, hepatic, or cardiopulmonary functions.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events | 15days or 22days
Safety as assessed by temperature | 15days or 22days
Safety as assessed by systolic blood pressure, diastolic blood pressure | 15days or 22days
Safety as assessed by pulse rate | 15days or 22days
Safety assessed by physical findings examinations, including weight | 15days or 22days
Safety as assessed by Laboratory test values | 15days or 22days
  Laboratory tests include hematology, biochemistry, urine analysis and coagulation
Safety as assessed by ECGs | 15days or 22days
Plasma concentrations and PK parameters (AUC, Cmax, Tmax, total clearance, volume of distribution and T1/2) of PCO371 in healthy male volunteers | 15days or 22days
Urine concentrations and PK parameters (cumulative excretion and renal clearance) of PCO371 | 15days or 22days

SECONDARY OUTCOMES:
The Time profile of serum/plasma concentrations in albumin-corrected total calcium (Ca); 25-hydroxy vitamin D (vit D), 1,25-dihydroxy vit D, and 24,25-dihydroxy vit D; phosphate; magnesium; and cAMP of PCO371 | 15days
The Urinary excretion of Ca, phosphate, magnesium, protein, sodium, potassium, chloride, and cAMP of PCO371 | 15days
The Nephrogenous cAMP of PCO371 | 15days

CONTACTS AND LOCATIONS:
Overall Officials: Ger Rikken, Study Director — Chugai Pharmaceutical
Locations (1):
- Wcct Global, Cypress, California, United States